CLINICAL TRIAL: NCT00362193
Title: Longitudinal Diabetes Care: A Randomized Controlled Trial to Prevent Glycemic Relapse
Brief Title: Glycemic Relapse Prevention: Maintenance Dose Assessment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Vanderbilt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK62258 (completed); P60DK020593 (NIH)
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Chronic disease management; Relapse
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Recurrence

INTERVENTIONS:
Behavioral: Telephonic diabetes care

SUMMARY:
This purpose of this study is to determine the optimal frequency of maintenance intervention needed to prevent glycemic relapse.

DETAILED DESCRIPTION:
Recent large randomized controlled trials have proven that tight glycemic control reduces the microvascular and macrovascular complications of diabetes. Reduction of these complications also leads to a great cost savings to healthcare and society. However, it has been difficult to translate the success of these large randomized control trials to everyday practice. A recent cross-sectional analysis of 95 clinicians revealed only 40.5% of type 2 diabetes patients had a glycated hemoglobin (HbA1c) less than 7%. The disparity of care between the large trials and a primary care office is largely due to the difference in resources available in the typical medical office. Practical, sustainable ways of maintaining tight glycemic control are needed in everyday practice.

While diabetes improvement programs are successful in acutely lowering HbA1c the long-term effectiveness of these programs is disappointing. Approximately 40% of those who return to routine care after completing an intensive diabetes improvement program experience a relapse in their glycemic control within one year. Some proportion of the relapse is likely due to a patient's inability to maintain adherence to key self-care behaviors - diet, exercise, self-monitoring of blood glucose and medication regimen.

The purpose of this study is to better understand prevention of glycemic relapse. The primary aim of this study is to assess the relative effectiveness of three management approaches, varying in frequency, for preventing glycemic relapse after glycemic control has been achieved through participation in an intensive diabetes improvement program. This study will determine the optimal frequency of intervention needed to prevent glycemic relapse in patients with type 2 diabetes. The authors hypothesize that high intensity intervention will lead to a decrease in glycemic relapse in a dose dependent fashion.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Recent control obtain (HbA1c<8%) after diabetes improvement program
* Receives care in primary care clinic

Exclusion Criteria:

* pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165
Dates: Start 2002-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Glycemic relapse: increase in HbA1c by 1% over baseline and >8%

SECONDARY OUTCOMES:
Height/Weight
Waist/Hip Circumference
Systolic/Diastolic BP
Demographic variables
Duration of Diabetes (years)
Hypoglycemia
3-day food record
SF-36
Self Efficacy
Medication
Medication Adherence
Exercise
Self-monitoring blood glucose (obtained from DIP records)
Fasting Lipid Panel

CONTACTS AND LOCATIONS:
Overall Officials: Tom A Elasy, MD, MPH, Principal Investigator — Vanderbilt University

REFERENCES:
- [Derived] Huizinga MM, Gebretsadik T, Garcia Ulen C, Shintani AK, Michon SR, Shackleford LO, Wolff KL, Brown AW, Rothman RL, Elasy TA. Preventing glycaemic relapse in recently controlled type 2 diabetes patients: a randomised controlled trial. Diabetologia. 2010 May;53(5):832-9. doi: 10.1007/s00125-010-1658-3. Epub 2010 Jan 19. PMID 20084363